CLINICAL TRIAL: NCT04632615
Title: Sleep Behaviour in Athletes During Home Confinement Due to the Covid-19 Outbreak
Acronym: Sleep&Covid19
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: Sleep&Covid19
Record Dates: First submitted 2020-11-12; First posted 2020-11-17 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Sleep; Athlete; Training; Exercise; Covid19; Isolation, Social
MeSH Terms: conditions — Motor Activity; COVID-19; Social Isolation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is becoming increasingly evident that sleep plays an essential role for human health, and it represents an important biophysiological variable for athletes' well-being and recovery. The International Olympic Committee recently highlighted the importance of obtaining sufficient sleep volume and quality among athletes, but acute sleep deprivation is not unusual. Several factors, both endogenous and exogenous, are able to negatively influence sleep in athletes: body temperature, altitude, chronotype, training volume, anxiety, westward and eastward travels, and many others.

Since December 2019, when a new coronavirus (SARS-CoV-2) was originally revealed by an ophthalmologist in Wuhan (Hubei province, China), a related severe acute respiratory syndrome - namely COVID-19 - has been spreading at a pandemic rate, putting global health systems under unprecedent pressure. Italy, as the first Western country tremendously hit by this disease outbreak, has become the iconic resilient outpost under international policymakers' attention. When initial clusters were identified, restrictive actions to curb isolated upsurges of infection were taken by the health region system of Lombardy, thereafter, were extended to all northern Italy and to the entire country. From February 21, when the first Italian COVID-19 case was diagnosed in southern Lombardy, to March 22, when Italian's government restrictions to contain the pandemic were extended, prohibiting all non-essential business activities and banning all movements of people nationwide, the country faced an unchartered scenario, from several standpoints, along with the psychosocial one.

Inevitably, the Covid-19 outbreak has largely influenced the daily life of athletes too. Therefore, the primary aim of this study was to examine the differences in athletes' sleep quality, quantity and training volumes during the social confinement due to the virus outbreak. For this purpose, a survey will be used. This variables will be evaluated in 3 different time frames: 1) May 2020; 2) September 2020; 3) January 2021.

ELIGIBILITY:
Inclusion Criteria:

* male or female gender.
* age between 18 and 40 years old.
* elite athletes (competing at national or international level).
* no cognitive impairments.
* at least 6 years of practice of a specific sport discipline.
* affiliated to CONI (Comitato Olimpico Nazionale Italiano).

Exclusion Criteria:

* age under 18 years old.
* part-time workers.
* injury or any clinical condition affecting training routines (and sleep).
* pregnant women.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Italian elite athletes will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Subjective sleep quality | This outcome will be evaluated in 3 different time frames: 1) May 2020; 2) September 2020; 3) January 2021.
  Subjective sleep quality of athletes will be evaluated by the completion of a survey.
Change in Subjective sleep quantity | This outcome will be evaluated in 3 different time frames: 1) May 2020; 2) September 2020; 3) January 2021.
  Subjective sleep quantity of athletes will be evaluated by the completion of a survey.
Change in Training volume | This outcome will be evaluated in 3 different time frames: 1) May 2020; 2) September 2020; 3) January 2021.
  Athletes' weekly training volume will be evaluated by the completion of a survey.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Vitale KC, Owens R, Hopkins SR, Malhotra A. Sleep Hygiene for Optimizing Recovery in Athletes: Review and Recommendations. Int J Sports Med. 2019 Aug;40(8):535-543. doi: 10.1055/a-0905-3103. Epub 2019 Jul 9. PMID 31288293
- [Result] Vitale JA, Weydahl A. Chronotype, Physical Activity, and Sport Performance: A Systematic Review. Sports Med. 2017 Sep;47(9):1859-1868. doi: 10.1007/s40279-017-0741-z. PMID 28493061
- [Result] Vitale JA, Roveda E, Montaruli A, Galasso L, Weydahl A, Caumo A, Carandente F. Chronotype influences activity circadian rhythm and sleep: differences in sleep quality between weekdays and weekend. Chronobiol Int. 2015 Apr;32(3):405-15. doi: 10.3109/07420528.2014.986273. Epub 2014 Dec 3. PMID 25469597
- [Result] Vitale JA, La Torre A, Banfi G, Bonato M. Acute sleep hygiene strategy improves objective sleep latency following a late-evening soccer-specific training session: A randomized controlled trial. J Sports Sci. 2019 Dec;37(23):2711-2719. doi: 10.1080/02640414.2019.1661938. Epub 2019 Sep 6. PMID 31608830
- [Result] Vitale JA, Banfi G, Sias M, La Torre A. Athletes' rest-activity circadian rhythm differs in accordance with the sport discipline. Chronobiol Int. 2019 Apr;36(4):578-586. doi: 10.1080/07420528.2019.1569673. Epub 2019 Feb 14. PMID 30760036
- [Result] Pillay L, Janse van Rensburg DCC, Jansen van Rensburg A, Ramagole DA, Holtzhausen L, Dijkstra HP, Cronje T. Nowhere to hide: The significant impact of coronavirus disease 2019 (COVID-19) measures on elite and semi-elite South African athletes. J Sci Med Sport. 2020 Jul;23(7):670-679. doi: 10.1016/j.jsams.2020.05.016. Epub 2020 May 19. PMID 32448749
- [Result] Di Renzo L, Gualtieri P, Pivari F, Soldati L, Attina A, Cinelli G, Leggeri C, Caparello G, Barrea L, Scerbo F, Esposito E, De Lorenzo A. Eating habits and lifestyle changes during COVID-19 lockdown: an Italian survey. J Transl Med. 2020 Jun 8;18(1):229. doi: 10.1186/s12967-020-02399-5. PMID 32513197
- [Result] Hakansson A, Jonsson C, Kentta G. Psychological Distress and Problem Gambling in Elite Athletes during COVID-19 Restrictions-A Web Survey in Top Leagues of Three Sports during the Pandemic. Int J Environ Res Public Health. 2020 Sep 14;17(18):6693. doi: 10.3390/ijerph17186693. PMID 32937978